CLINICAL TRIAL: NCT01689220
Title: A Phase 1 Study of SP-02L (Darinaparsin for Injection) in Relapsed or Refractory Patients With Peripheral T-cell Lymphoma (PTCL) in Korea
Brief Title: A Phase 1 Study of SP-02L in Relapsed or Refractory Patients With Peripheral T-cell Lymphoma (PTCL) in Korea
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Solasia Pharma K.K. (Industry)
Collaborators: Synex Consulting Korea Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP-02L03
Record Dates: First submitted 2012-09-14; First posted 2012-09-21 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-09

CONDITIONS: Peripheral T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — darinaparsin; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SP-02L (Experimental)
  Interventions: Drug: SP-02L (darinaparsin for injection)

INTERVENTIONS:
Drug: SP-02L (darinaparsin for injection) — Cohort 1: Darinaparsin 300 mg/m2 for 5 consecutive days every 28 days (5 days therapy, 23 days no therapy is one cycle). Subjects may start from Cycle 1 and continue to a maximum of 4 cycles of treatment.
Drug: SP-02L (darinaparsin for injection) — Cohort 2: Darinaparsin 300 mg/m2 for 5 consecutive days every 21 days (5 days therapy, 16 days no therapy is one cycle). Subjects may start from Cycle 1 and continue to a maximum of 4 cycles of treatment.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of SP-02L monotherapy in Korean patients with relapsed or refractory Peripheral T-cell Lymphoma (PTCL).

ELIGIBILITY:
Inclusion Criteria:

* Korean patients aged ≥ 20 years of age at the day of obtaining the informed consent
* Patients with histologically confirmed diagnosis of the following:

  * PTCL, not otherwise specified (PTCL-NOS)
  * Anaplastic Large Cell Lymphoma (ALCL ALK-positive/negative)
  * Angioimmunoblastic T-cell Lymphoma (AITL)
* Have relapsed or refractory to at least one prior systemic chemotherapy for the above disease (currently requiring therapy)
* Have at least 1 evaluable lesion
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Life expectancy of at least 3 months

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-09; Primary Completion 2014-01 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity and adverse events | 12 or 16 weeks

SECONDARY OUTCOMES:
Tumor response (overall response) | 2 and 4 cycles
Plasma concentration-time profile | 0, 0.5, 1, 2, 4, 8 hours post-dose on Day 1 and 5, and 0 hour on Day 2, 3, 4, 6, 8 and 15
  Cmax, Area under curve, Tmax, t1/2, Clearance and Volume of distribution

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Ogura M, Kim WS, Uchida T, Uike N, Suehiro Y, Ishizawa K, Nagai H, Nagahama F, Sonehara Y, Tobinai K. Phase I studies of darinaparsin in patients with relapsed or refractory peripheral T-cell lymphoma: a pooled analysis of two phase I studies conducted in Japan and Korea. Jpn J Clin Oncol. 2021 Feb 8;51(2):218-227. doi: 10.1093/jjco/hyaa177. PMID 33051668